CLINICAL TRIAL: NCT03189758
Title: Dietary Sodium (DS) Intervention to Reduce Volume Overload and Tissue Sodium in Magnetic Resonance Imaging (MRI) for Hemodialysis (HD) Patients
Acronym: DSMRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Renal Research Institute (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 17530
Record Dates: First submitted 2017-06-14; First posted 2017-06-16 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Kidney Failure, Chronic; Dietary Modification
Keywords: chronic kidney disease; hemodialysis; sodium restriction; MRI
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Observational control followed by dietary intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Participants will follow a Observational Control Diet (CON) diet followed by an Controlled Dietary Sodium Restriction (INT) diet.
  Interventions: Other: Observational Control Diet; Other: Controlled Dietary Sodium Restriction

INTERVENTIONS:
Other: Observational Control Diet — Participants will follow their usual or normal diet for 30 days (days 1-30) while under study observation.
  Other Names: CON
Other: Controlled Dietary Sodium Restriction — Participants will be provided with all meals and snacks daily, for 30 days (days 31-60). These meals should meet KDQOI guidelines for energy and protein (30-35 kcal/kg & 1.2 g/kg) as well as low phosphorus, potassium, and sodium. The meals are formulated to less than 600-800 mg sodium each (<2,000g/day) and will be ordered and delivered through momsmeals.com
  Other Names: INT

SUMMARY:
Sodium-adapted magnetic resonance imaging (23Na-MRI) studies have demonstrated that sodium accumulates in certain tissues, including the skin and skeletal muscle, but may be manipulated by lifestyle factors or therapeutic interventions such as a hemodialysis (HD) session. This tissue sodium accumulation is increased with age and in the presence of certain chronic diseases such as renal failure, and may contribute to the development of high blood pressure. It currently not known what the impact of dietary sodium consumption has on tissue sodium in HD patient's and on the subsequent risk of cardiovascular complications either acutely or chronically. The University of Illinois' Biomedical Imaging Center recently completed safety testing on a 23Na-MRI coil that they modified for measuring skin and muscle sodium levels in the lower leg/calf that will be used for assessing the impact of dietary salt restriction on tissue sodium levels.

DETAILED DESCRIPTION:
Recent studies illustrate that tissue sodium is regulated by immune cells in interstitial fluids such as the skin and muscle. Localized immune responses in these tissues can promote vascular endothelial growth factor secretion to promote lymphatic release of fluid and electrolytes, which has significant implications for blood pressure control and cardiovascular health. Furthermore, sodium composition of the diet has the potential to promote beneficial gut bacteria in addition to lowering auto-immune response and blood pressure.

The purpose of this pilot study is to utilize this 21Na-MRI coil to quantify changes of sodium levels in the skin and skeletal muscle in hemodialysis treatments before and after a low-sodium diet intervention. In this study, all HD patients will undergo a 30-day observation period (CON) followed by a low-sodium diet period (INT) for 30 additional days. Testing will occur at baseline and after each time-point (three time points total). During the CON period, patients will have no changes to their normal dialysis treatment, and will be asked to follow their normal diet. During the INT period, patients will provided a low- sodium diet intervention that includes receiving 3 low sodium meals per day and snacks provided by momsmeals.com.

The study outcomes include: clinical outcomes (hospitalizations, treatment efficiency) changes in tissue sodium, cardiovascular measures (blood pressure, cardiac output, and vascular resistance) and fluid/hydration status (total body water, extracellular fluid) using bioelectrical impedance. We will also collect serum to analyze the relationship between changes in tissue sodium and serum minerals (e.g. sodium and potassium), and other factors believed to help regulate tissue sodium levels, including vascular endothelial growth factor (VEGF), and markers of inflammation (CRP, IL-6). Additionally, we plan to collect patient stool samples to analyze how changes in dietary sodium consumption impact the gut microbiome.

This study will demonstrate the feasibility of utilizing 23Na-MRI to quantify skin and muscle sodium levels, as well as provide pilot data regarding the relationship between tissue sodium accumulation, inflammation, the gut microbiome, insulin resistance, and cardiovascular health in hemodialysis patients. Results from this study will then be used to design larger trials to investigate related questions.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to sign informed consent document and age 18 or greater.
* Willingness to consume intervention meals 3 times per day (with provided snacks) for 30 days.

Exclusion Criteria:

1. Individuals with pacemakers (exclusion from cardiovascular testing only)
2. Individuals with major amputations (i.e. whole limb: foot, ankle, leg, arm)
3. Individuals with ferric metal implants or devices in the body (excluded from MRI testing only)
4. Claustrophobic individuals (excluded from MRI testing only)
5. Individuals that do not otherwise meet MRI screening requirements (mentioned below, excluded from MRI testing only)
6. Individuals on HD therapy <3 days per week or <3 months
7. Currently following a sodium restricted diet approximately <1,500 mg per day (only excluded from MRI analysis)
8. Currently diagnosed GI disorder or disease or infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-06-19 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Interdialytic weight gain | 28 days
  Interdialytic weight from clinic records
Tissue sodium | 28 days
  MRI detected sodium content in the lower leg (mM)

SECONDARY OUTCOMES:
Hydration status | 28 days
  Bio-impedance measured total body water, extracellular fluid, intracellular fluid, and calculated fluid volume overload
Cardiovascular function | 28 days
  Standard blood pressure
Biochemical markers | 28 days
  Vascular endothelial growth factor-C (VEGF-C), C-reactive protein (CRP), interleukin (IL-6), tumour necrosis factor alpha (TNF-a), endothelial nitric oxide (eNOS), serum sodium (Na)
Gut microbiome (stool sample) | 28 days
  DNA sequencing, bacteria phyla and taxa, stool consistency, gastrointestinal symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided